CLINICAL TRIAL: NCT02239497
Title: Femoral Preincisional Block in Acute Postoperative Pain Management of Surgery Orthopaedic Lower Limb
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Central Dr. Luis Ortega (Other)
Responsible Party: Principal Investigator, Beatriz Arismendi Gómez, Anesthesiologist, Hospital Central Dr. Luis Ortega
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Femoral Block
Record Dates: First submitted 2014-09-07; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Surgery
Keywords: postoperatory pain; orthopaedic surgery; femoral block

ARMS (2):
- femoral block by US and NE and intravenous analgesia (Experimental): preincisional femoral block by ultrasound and neurostimulation, with 20 ml bupivacaine 0,5% and epinephrine. ketoprofen, dipyrone and dexamethasone IV. Morphine IV to rescue analgesia
  Interventions: Procedure: Femoral block by ultrasound and neurostimulation; Drug: Intravenous analgesia
- Intravenous analgesia (Experimental): Intravenous analgesia with ketoprofen, dipyrone and morphine. IV morphine to rescue analgesia
  Interventions: Drug: Intravenous analgesia

INTERVENTIONS:
Procedure: Femoral block by ultrasound and neurostimulation
  Arms: femoral block by US and NE and intravenous analgesia
Drug: Intravenous analgesia — Intravenous analgesia with ketoprofen, dipyrone and dexamethasone. IV morphine to rescue analgesia

SUMMARY:
Proper management of acute postoperative pain (DAPO) is essential for the recovery of orthopedic surgeries. The blockade of the femoral nerve preincisional (BFP) is simple and its effectiveness increases guided by ultrasound and neurostimulation. OBJECTIVE: To evaluate the effectiveness of BFP in patients undergoing orthopedic surgery of the lower limbs under general anesthesia. METHODS: A comparative study was conducted, randomized, two groups, surgeries of the hip, femur and knee, ASA I-II, aged 18 years. Group B (n = 15) received BFP and ultrasound-guided nerve stimulation with 20 ml of bupivacaine 0.5% plus epinephrine 1: 200,000. Group S (n = 15) without blocking. Both groups received intravenous analgesia with ketoprofen 100 mg regimen and dipyrone 1g c / 8 hs and balanced general anesthesia. Postoperative morphine 0.03 mgr / kgr / weight was administered if EVA ≥4

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients, both sexes, plan for elective orthopaedic surgery of the lower limbs (femur and knee) under general anesthesia

Exclusion Criteria:

* Patients with any anesthetic or surgical complication
* Patients with neuromuscular diseases
* Allergy to any of the drugs used in the study
* Inability to understand and use a pain scale
* Also those patients in whom it was not possible to locate anatomical landmarks and / or failed femoral block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Postoperatory EVA values and need for rescue analgesia with IV morphine | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz S Arismendi Gomez, MD, Principal Investigator — Hospital "Dr Luis Ortega"
Locations (1):
- Servicio de Anestesiologia Hospital "Dr. Luis Ortega", Porlamar, Nueva Esparta, Venezuela